CLINICAL TRIAL: NCT02264912
Title: The Laboratory AntiPlatelet Efficacy and Clinical Outcome Registry
Acronym: LAPCOR
Status: Completed | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Zuzana Motovska, Associate Professor, MD. PhD. FESC., Faculty Hospital Kralovske Vinohrady
Other Study IDs: 05-2008
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Platelet Aggregation Onhibitors
Keywords: antiplatelets, percutanous coronary intervention, acute coronary syndromes, laboratory efficacy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stent-PCI patients: Consecutive patients, who underwent intracoronary stent implantation, have been included regardless of whether percutaneous coronary intervention (PCI) was performed on urgent or elective basis.
  Interventions: Drug: antiplatelet drugs - P2Y12 antagonists

INTERVENTIONS:
Drug: antiplatelet drugs - P2Y12 antagonists
  Other Names: clopidogrel, prasugrel, ticagrelor

SUMMARY:
The ongoing LAPCOR (Laboratory AntiPlatelet efficacy and Clinical Outcome Registry) registry was initiated in 2008 at a tertiary care cardiac center, and consecutive patients, who underwent intracoronary stent implantation, have been included regardless of whether percutaneous coronary intervention (PCI) was performed on urgent or elective basis.Patients were included in the registry after having signed an informed consent for participation. No exclusion criterion has been applied for the registry participation. Efficacy of P2Y12 receptor antagonists has been measured by quantitative flow cytometric analysis of vasodilator-stimulated phosphoprotein (VASP) phosphorylation according to the manufacturer protocol (Platelet VASP; Diagnostica Stago, Biocytex, Asnières, France) on a FACScan flow cytometer (Becton Dickinson). Occurrence of major adverse cardiac events at 30 days, 6-months and one year follow up has been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients after stent PCI treated with P2Y12 antagonist
* Written informed consent

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included in the registry after having signed an informed consent for participation. No exclusion criterion has been applied for the registry participation.
Sampling Method: Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2008-07; Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
laboratory efficacy of antiplatelet drugs measured as residual platelet reactivity, incidence of major adverse cardiovascular events and bleeding complications | During the 12 months after implantation of an intracoronary stent

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Motovska, MD.PhD., Principal Investigator — Faculty Hospital Kralovske Vinohrady
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

REFERENCES:
- [Result] Motovska Z, Odvodyova D, Fischerova M, Stepankova S, Maly M, Morawska P, Widimsky P. Renal function assessed using cystatin C and antiplatelet efficacy of clopidogrel assessed using the vasodilator-stimulated phosphoprotein index in patients having percutaneous coronary intervention. Am J Cardiol. 2012 Mar 1;109(5):620-3. doi: 10.1016/j.amjcard.2011.10.019. Epub 2011 Dec 10. PMID 22154314
- [Result] Motovska Z, Ondrakova M, Doktorova M, Widimsky P. Severe left ventricular systolic dysfunction is independently associated with high on-clopidogrel platelet reactivity. Am J Cardiovasc Drugs. 2014 Aug;14(4):313-8. doi: 10.1007/s40256-014-0074-3. PMID 24728851
- [Result] Ondrakova M, Knot J, Ulman J, Maly M, Motovska Z. Efficacy of P2Y12 receptor antagonists in patients with atrial fibrillation according to the CHA2DS2VASc score. Int J Cardiol. 2016 Mar 15;207:84-6. doi: 10.1016/j.ijcard.2016.01.039. Epub 2016 Jan 6. No abstract available. PMID 26797336
- [Result] Motovska Z, Ondrakova M, Bednar F, Knot J, Ulman J, Maly M. Selection of P2Y12 antagonist, treatment initiation, and predictors of high on-treatment platelet reactivity in a "Real World" registry. Thromb Res. 2015 Jun;135(6):1093-9. doi: 10.1016/j.thromres.2015.04.014. Epub 2015 Apr 16. PMID 25917561